CLINICAL TRIAL: NCT02444052
Title: Clinical and Histological Evaluation of Zimmer Puros® Allograft vs. Creos™ (Low-cost) Allograft for Alveolar Ridge Preservation Following Exodontia
Brief Title: Evaluation of Zimmer Puros® Allograft vs. Creos™ Allograft for Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20150016
Record Dates: First submitted 2015-05-07; First posted 2015-05-14 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Alveolar Bone Grafting; Allograft; Dental Extraction; Dental Implant; Socket Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zimmer Puros Cancellous Allograft (Experimental): Right side will have an extraction followed by an allogenic bone graft zimmer puros followed by implant placement.
  Interventions: Device: Zimmer Puros Cancellous Allograft
- Nobel Biocare Creos Cancellous Allograft (Experimental): Left side will have an extraction followed by an allogenic bone nobel biocare creos graft followed by implant placement.
  Interventions: Device: Nobel Biocare Creos Cancellous Allograft

INTERVENTIONS:
Device: Zimmer Puros Cancellous Allograft — Right side will have an extraction followed by an allogenic bone graft zimmer puros followed by implant placement.
  Arms: Zimmer Puros Cancellous Allograft
Device: Nobel Biocare Creos Cancellous Allograft — Left side will have an extraction followed by an allogenic bone nobel biocare creos graft followed by implant placement.
  Arms: Nobel Biocare Creos Cancellous Allograft

SUMMARY:
The purpose of this study is to evaluate clinically, histologically and radiographically the healing of extraction sockets with Zimmer's Puros® allograft compared to creos™ (creo™ Nobel Biocare,), a low-cost allograft material, 90 days following exodontia.

DETAILED DESCRIPTION:
Twenty-four consecutive subjects requiring extraction of two non-adjacent molars or premolars located in the same jaw will be selected from the patient pool of the Center for Advanced Periodontology at the University of Florida, College of Dentistry.

Preoperative Procedures: At the initial screening, the goals of the study, potential risks and possible benefits will be explained and each subject will be asked to sign a written consent statement permitting extraction of the involved teeth and the placement of Puros® allograft and creos™ allograft for ridge preservation. After which a complete medical and dental history will be obtained, a pregnancy test will be performed, and establishment of inclusion and exclusion criteria will be determined. If meeting all study criteria, examination periapical radiographs will be taken and each subject will receive oral hygiene instructions, prophylaxis, and full-arch alginate impressions. The study models will also be used to fabricate occlusal templates to permit reproducible clinical measurements of the alveolar ridge dimensions of the residual tooth socket.

Surgical Protocol & Treatment Assessment: To help minimize technical variances in the surgical treatment protocol, the primary investigator will perform baseline and 12-week re-entry surgeries. Under local anesthesia, full-thickness mucoperiosteal flaps will be elevated; the selected teeth will be extracted atraumatically, followed by debridement of the sockets, and collection of all clinical measurements.The following clinical measurements will be made at the baseline and re-entry surgeries using standard University of North Carolina (UNC) manual probes (Hu-Friedy, Chicago, IL):

1. Facial/buccal thickness (baseline, only)
2. Distance from the occlusal template to the facial, lingual and crestal bone
3. Socket depth (or template to crest distance at the 90-day re-entry surgery)
4. Osseous dehiscence location and dimension
5. Bone density (on re-entry)

The surgeon will then preserve each site with either Puros® allograft creos™ allograft. Puros® allograft will be placed into half of the extraction sockets to the level of the osseous crest. A bovine pericardium membrane (CopiOs ®Pericardium) will be then placed to cover the bone graft material. Primary closure will be achieved in all cases. The site will be sutured with 4.0 PTFE sutures. The other extraction sites will receive the same treatment but with creos™ allograft. Participants will be prescribed a 10 day regimen of Ibuprofen (2.4g/day) and antibiotics (amoxicillin (1.5g/day) or clindamycin (0.6g/day)) unless other allergies are present. Subjects will be instructed to change their diet to semi-liquid for 48 hours, followed by soft foods for the first 2-weeks. Subjects will also be instructed to begin rinsing with warm water, as needed, and to resume their normal oral hygiene routine the day after surgery in all areas except the surgical site.

At 2-week post-surgery, the extraction sites will be inspected and gently cleaned with saline-soaked gauze, health histories will be reviewed, oral hygiene instructions will be repeated, photographs will be taken; and a plaque score will be recorded. Cone beam CT images will be performed 2 weeks and 12 weeks post-operative. All imaging will be done using the Kodak limited view CBCT to minimize the subjects' exposure to radiation.

Soft tissue healing will be assessed at 2, 8 and 12 weeks with a wound-healing index (WHI) according to the following scheme: score "1" for uneventful wound healing with no gingival edema, erythema, suppuration, discomfort or graft exposure; score "2" for uneventful wound healing with slight gingival edema, erythema, or discomfort, but minimal loss of graft and no suppuration; score "3" for poor wound healing with significant gingival edema, erythema, discomfort, loss of graft or any suppuration.

Re-entry surgery will be performed at 12 weeks, and all clinical measurements will be repeated. Crestal flapless soft tissue and bone core biopsies approximately 2.7 x 10 mm in size will be removed with a 3.2 mm trephine drill from the area corresponding to the center of the previous extraction from the crest of the ridge using the occlusal template as a guide.

The cores will be placed in bottles of 10% neutral buffered formalin (NBF) for fixation, and then labeled with a 5-digit number in order to permit masked histomorphometric analysis. Analysis will be performed in the outer aspect of the bone cores, which correspond to the bone surface that will contact the dental implants at the time of placement. Zimmer TSTV implants will be placed at the same time the second re-entry procedure is done. All implants will be placed according to the manufacturer's specifications. Restorative treatment will be initiated 90 days after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects with two non-adjacent molar or premolar teeth located in the same jaw that require extraction and socket augmentation for implant site development (treatment sites may be located in either the mandibular or maxillary jaw)
* Residual extraction sockets must have <70% bone loss in all dimensions (3 or 4-walled bony defects)
* Nonsmokers (individuals who quit smoking at least 6 months prior to the study will be allowed to participate)
* Subjects willing and able to comply with all study-related procedures including maintenance of good oral hygiene and compliance with re-evaluation appointments
* Subjects who read, understand and are willing to sign an informed consent statement.

Exclusion Criteria:

* Inadequate zone of keratinized gingiva (KG) or alveolar mucosa to obtain primary wound closure of the surgical site
* Presence of acute infections at the time of tooth extraction
* Clinically significant or unstable (as defined by the investigators) systemic diseases affecting bone or soft tissue growth; or other renal, hepatic, cardiac, endocrine, hematologic, autoimmune or acute infectious diseases that makes interpretation of the data more difficult
* History of head & neck radiation therapy
* Subjects taking steroids, tetracycline or tetracycline analogs, bone therapeutic levels of fluorides, biphosphonates, medications affecting bone turnover, antibiotics for >7 days or any investigational drug
* Patients who are or become pregnant during the length of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Bone change in millimeters from initial (baseline) to full healing (week 12) | At week 12
Cone beam computed tomography bone density changes | At week 12
Percentage of bone formation in the alveolar bone core biopsies | At week 12
Percentage of volumetric bone formation observed by comparison of Cone beam computed tomography images and the percentage of residual Puros® bone cores | At week 12
Percentage of volumetric bone formation observed by comparison of Cone beam computed tomography images and the percentage of residual creos™ allograft in the bone cores | At week 12

SECONDARY OUTCOMES:
Facial/buccal alveolar bone thickness measured in millimeters with calipers | At Baseline
  After extraction of the tooth, the facial/buccal bone thickness will be measured with calipers to the nearest millimeter.
Length of alveolar dehiscence defects measured in millimeters with a periodontal probe | At Baseline
  This measurement is made after the tooth is extracted and measured with a periodontal probe to the nearest millimeter
Width of alveolar dehiscence defects measured in millimeters with a periodontal probe | At Baseline
  This measurement is made after the tooth is extracted and measured with a periodontal probe to the nearest millimeter
Plaque score | Pre-op, Baseline, Week 2, 8 and 12
  A disclosing solution such is painted on all exposed tooth surfaces. After the patient has rinsed, the operator (using an explorer or a tip of a probe) examines each stained surface for soft accumulations at the dentogingival junction. When found, they are recorded by making a dash/red color in the appropriate spaces on the record form. Those surfaces, which do not have soft accumulations at the dentogingival junction, are not recorded.
Subjective clinical bone density on re-entry | At week 12
  Assessed during osteotomy for implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Neiva, DDS,MS, Principal Investigator — Program Director Grad Perio UFCD
Locations (1):
- University of Florida College of Dentistry-Periodontics, Gainesville, Florida, United States